CLINICAL TRIAL: NCT05669157
Title: X-rays Trauma Request's by the Triage And Intake Nurse Intake and Referral Nurse: X-TRAIN Study
Brief Title: X-rays Trauma Request's by the Triage And Intake Nurse Intake and Referral Nurse:
Acronym: DARIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHRO-2022-08
Record Dates: First submitted 2022-12-12; First posted 2022-12-30 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Limb Injury
Keywords: Traumatology; Personnel delegation; Nurse specialists; Radiography; emergency department; intake and referral nurse
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current practice: radiography request by physician (Experimental): No interventions will be performed. There is no change in current practice.
  Interventions: Procedure: Radiography request by physician
- Radiography request by the nurse (Experimental): the intake and referral nurse will request a radiography if required according to the local cooperation protocol
  Interventions: Procedure: Radiography request by nurse

INTERVENTIONS:
Procedure: Radiography request by nurse — Intervention group with radiography requested by the IRN instead of the physician. The radiography will be interpreted by the physician afterwards, according to current practice
  Arms: Radiography request by the nurse
Procedure: Radiography request by physician — The physician prescribed the X-ray, the X-ray technician carries out the imagery and the physician interprets it afterwards
  Arms: Current practice: radiography request by physician

SUMMARY:
The number of consultations in emergency departments is increasing day by day, and the time to treat patients is getting longer. Different French studies have shown a significant reduction in the time spent in the emergency department after the implementation of the national protocol for the delegation of early radiography prescriptions. The investigators hypothesised that an early request for a standard X-ray by the intake and referral nurse in the case of isolated trauma to the extremities of a limb (from the knee to the toes and from the shoulder to the fingers) enables a reduction in medical management time and, consequently, in the time spent in the emergency department for the patient.

DETAILED DESCRIPTION:
This study is divided into two steps to three month.

* The first step of the study corresponds to the current standard of care (SoC) in the emergency department of Orléans. In this first step, the intake and Referral Nurse (IRN) will carry out the usual triage and refer the participant to the appropriate emergency department before being appointed by the physician. The radiography will be requested after the medical consultation.
* In the second step, the intake and referral nurse will carry out the usual triage and then request one, or more, radiography(ies) depending on the standard protocol. This ensures that the physician has access to the imaging before the consultation with the patient. If necessary, the X-ray technician is authorized to refuse the exams or complete the request, the choice of the incidence is up to him/her according to the intake and referral nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 15 years and 3 months admitted in adult emergency department of regional hospital center of ORLEANS with a simple and isolated trauma having occurred less than 48 hours prior to admission of a limb extremity (from the knee to the toes or from the shoulder to the fingers), and with no previous imagery assessment within 48 hours prior to admission in the emergency department.

Exclusion Criteria:

* Multiple trauma
* Patient with at least one Vittel criteria (except age)
* Patient refusing the protocol
* Hemodynamic instability and/or disorder of consciousness
* Sensory and/or vascular disorders downstream of the traumatized area
* Protected population (under guardianship or curators)
* Patient under court protection
* Pregnant or breastfeeding woman or one who declares herself to be pregnant or breastfeeding
* Patient with an expired blood alcohol level > 0.4 mg/L and/or positive blood alcohol level
* Patient with diagnosed dementia
* Patient hospitalized after being taken in charge

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Duration between triage and exit of emergency unit | immediatly after the procedure
  Total duration in minutes in the emergency department with or without anticipated request of X-ray

SECONDARY OUTCOMES:
Total duration of the stay | immediatly after the procedure
  Total duration in minutes in the emergency department
Number of additional X-ray prescribed by the physician after physician assessment. | immediatly after the procedure
  Number of new X-ray images taken after physician assessment.
Appropriateness of the X-rays requested by the IRN as per guidelines | immediatly after the procedure
  Number of new X-ray images taken after physician assessment.
IRN's feeling about the anticipated request for X-ray (assessed as per anonym Quality of Life at Work questionnaire) | immediatly after the procedure
  Quality of life questionnaire. Min: not satisfied; max : satisfied
X-ray technician's feeling about the anticipated request for X-ray (assessed as per anonym Quality of Life at Work questionnaire) | immediatly after the procedure
  Quality of life questionnaire. Min: not satisfied; max : satisfied
Physician's feeling about the anticipated request for X-ray (assessed as per anonym Quality of Life at Work questionnaire) Physician's feeling about the anticipated request for X-ray (assessed as per anonym Quality of Life at Work questionnaire) | immediatly after the procedure
  Quality of life questionnaire. Min: not satisfied; max : satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GARROUSTE, MD, Principal Investigator — Regional Hospital center of ORLEANS
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindley-Jones M, Finlayson BJ. Triage nurse requested x rays--are they worthwhile? J Accid Emerg Med. 2000 Mar;17(2):103-7. doi: 10.1136/emj.17.2.103. PMID 10718230